CLINICAL TRIAL: NCT03228550
Title: Investigating the Effects of Omega-3 Fatty Acid Multinutrient Supplement and Exercise on Mobility and Cognition in Older Women
Brief Title: Omega-3 Fatty Acids and Exercise on Mobility and Cognition in Older Women
Acronym: MOBILE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: Efamol Ltd (Industry); Sylvia Waddilove Foundation (Unknown)
Responsible Party: Principal Investigator, Simon Dyall, Principal Academic, Bournemouth University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 002
Record Dates: First submitted 2017-07-10; First posted 2017-07-25 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Aging; Cognitive Decline
Keywords: omega-3 fatty acid; B vitamins; vitamin E; Phosphatidylserine; Gingko biloba; Gait; Aerobic Exercise; Memory; Cognitive function
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: There are two interventions, a multi-nutrient dietary supplement and exercise. The study will have four groups; 1. multi-nutrient supplement and exercise, 2. multi-nutrient non-exercise, 3. placebo supplement and exercise and 4. placebo supplement non-exercise.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants blinded to dietary intervention, but not exercise. Outcomes assessor blinded to both intervention and exercise group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Efamol Active 50+ and exercise (Experimental): Efamol Active 50+ Multinutrient supplement and aerobic exercise
  Interventions: Dietary Supplement: Efamol Active 50+; Behavioral: Aerobic exercise
- Efamol Active 50+ and non-exercise (Experimental): Efamol Active 50+ Multinutrient supplement and non-aerobic exercise
  Interventions: Dietary Supplement: Efamol Active 50+
- Placebo and exercise (Experimental): Placebo supplement and aerobic exercise
  Interventions: Behavioral: Aerobic exercise; Dietary Supplement: Placebo multinutrient
- Placebo and non-exercise (Experimental): Placebo supplement and non- exercise
  Interventions: Dietary Supplement: Placebo multinutrient

INTERVENTIONS:
Dietary Supplement: Efamol Active 50+ — 1000 mg docosahexaenoic acid, 160 mg eicosapentaenoic acid, 20 µg B12, 1 mg folic acid, 124 mg phosphatidylserine, 240 mg ginkgo biloba standardized leaf extract and 20 mg vitamin E
  Arms: Efamol Active 50+ and exercise; Efamol Active 50+ and non-exercise
Behavioral: Aerobic exercise — Static exercise cycle
  Arms: Efamol Active 50+ and exercise; Placebo and exercise
Dietary Supplement: Placebo multinutrient — Placebo multinutrient supplement
  Arms: Placebo and exercise; Placebo and non-exercise

SUMMARY:
The study will provide insight into how lifestyle-related interventions, specifically nutrition and exercise can impact the health of older women. The study uses a unique combination of interventions and encapsulates overall health outcomes by measuring both mobility and cognitive function.

The study examines the effects of a combined omega-3 polyunsaturated fatty acid (PUFA) and multi-nutrient supplement on measures of mobility and cognition in women aged 60 years and above. Volunteers for the study will be randomly assigned to one of four groups which are as follows:

* Omega-3 PUFA multi-nutrient supplement and aerobic exercise
* Omega-3 PUFA multi-nutrient supplement and no exercise
* Placebo supplement and aerobic exercise
* Placebo supplement and no exercise

Volunteers undertake the dietary supplementation for a period of 24 weeks. The active dietary supplement contains a daily dosage of 1 g docosahexaenoic acid, 160 mg eicosapentaenoic acid, 240 mg Ginkgo biloba, 60 mg phosphatidylserine, 20 mg d-α tocopherol, 1 mg folic acid, and 20 µg vitamin B12. The placebo supplement contains an iso-calorific oil blend that is typical of the current UK diet. The aerobic exercise consists of two classes per week the final 12 weeks of the study on stationary spinning exercise bikes.

Volunteers attend testing at the beginning and after 24 weeks. Verbal memory, spatial working memory, executive function and processing speed are assessed via a battery of cognitive tests. Mobility testing comprises three walking tests, some under single and dual task paradigms, as well as the five times sit to stand test, a measure of dynamic balance and functional mobility. Volunteers also provide two blood samples, one for fatty acids analysis and the other serum homocysteine levels. Participants also complete health-related quality of life questionnaire, the short form 36 (SF36) questionnaire, food diary and food frequency questionnaire.

DETAILED DESCRIPTION:
Design and Setting:

The study is a randomized semi-blinded, placebo-controlled trial in females aged 60 years and over. The study examines the effects of a high docosahexaenoic acid omega-3 PUFA multi-nutrient dietary supplement and aerobic exercise, both on their own and in combination, on outcomes related to mobility and cognition. All measurements and data collection, as well as the aerobic exercise, take place at the same study site (Bournemouth University, United Kingdom), with participants instructed to consume the dietary supplement at home.

Blinding Randomization and Allocation:

The dietary supplements are packed in identical containers and coded by the Principal Investigator, who has no involvement in the data collection. Omega-3 PUFA capsules have a distinct odor, therefore a small amount of fish oil is added to the placebo capsules to help maintain blinding. A stratified block randomization design is followed with stratification based on frailty classification of non-frail or pre-frail, followed by permuted block randomization. Randomization is achieved by creating a computer-generated list of numbers consisting of four blocks for each stratum referred to without specification of the intervention group (e.g., A, B, C, and D). The list is generated and stored by the Principal Investigator. Due to the nature of the exercise intervention participants are only be blinded to the dietary intervention; however, the experimenters are blinded to the exercise group allocations.

Participants:

Participants are recruited through local newspaper advertisements and public engagements in Bournemouth, U.K. The public advertisements include a brief study description as well as the contact details for the research team. Those who are interested receive a participant information document including the design, procedure, benefits, and risks of the study. Before any data is collected, all participants provide signed written informed consent forms.

All participants are screened to assess frailty status, according to the Fried et al. (2001) criteria. The criteria include low muscle strength, self-reported exhaustion, slowed gait speed, low levels of physical activity, and unintentional weight loss. A score of zero out of the five indicates non-frail, one or two pre-frail, and three or above frail.

The Mini Mental State Examination (MMSE) is performed to exclude participants with cognitive impairment, as this has the potential to go undiagnosed. The test is performed according to British Psychology Society guidelines, and is not used for diagnostic purposes and individual results are not be disclosed to any participant. Participants who score ≤24 are excluded from the study.

Demographic Information:

Information on the age, height, weight, verbal intelligence and medication use is collected from each participant. Information on medications is self-reported, with both type and number of medications recorded. The national adult reading test (NART) is used to assess verbal intelligence. The test requires participants to read aloud 50 pre-prepared words, with scores being calculated based on the number of correct pronunciations. Minor variations from the pronunciations are not penalized as the aim of the test is to assess familiarity with the words rather than exact pronunciation.

Sample Size:

Sample size was determined based on the primary outcome of habitual gait speed. The sample size calculation was based on a difference of 0.08 m/sec with a power of 0.8 and α of 0.05 (two-tailed), based on previous research (Strike et al. 2016). A minimum sample size of 25 participants per group is required to detect an effect size d of 0.8 between experimental groups and the control. An overall recruitment target of 120 participants, 30 per group has been set to allow for drop-outs.

Analysis will be carried out on the basis of groups as randomly assigned. This intention-to-treat analysis will include participants who decide to discontinue treatment, but take part in assessment at 24 weeks. Data analysis will be performed at the conclusion of the intervention and include data collected at baseline and 24 weeks. Data will be tested for normal distribution using Shapiro-Wilk test and Q-Q-plots. Associations between baseline levels of serum homocysteine, whole-blood DHA levels and cognitive and mobility outcomes will be made, as well as changes in DHA and measures of mobility and cognition at the end of the intervention. The treatment effects of the two interventions over time (from pre- and post-measurements) will be analyzed by 2 X 2 ANOVA, with demographic and health information, such as age and NART score, and changes in serum homocysteine and changes in blood fatty acids examined as covariates. This analysis will be performed on all primary and secondary outcomes. Effect size will also be calculated. In all analyses P<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk 50 meters unassisted
* Non-frail or pre-frail according to Fried frailty phenotype

Exclusion Criteria:

* Vestibular impairments
* Diagnosed neurological disorder
* Mini mental state examination score of ≤24
* History of lower limb surgery
* Seafood allergy
* Regular consumption of multivitamin/fish oil supplements within six months prior to baseline measurements
* Previously received advice from a health care professional to not take part in strenuous exercise.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Actual)
Dates: Start 2017-02-26 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in habitual gait speed | Baseline and 24 weeks post intervention
  Habitual gait speed will be measured using inertial measurement sensors and will be expressed in m/s. Participants will be asked to walk at their normal habitual pace over 13 m. Acceleration and deceleration periods will automatically be excluded from analysis and the measure will be repeated five times with the mean value calculated.

SECONDARY OUTCOMES:
Change in executive function | Baseline and 24 weeks post intervention
  Participants draw lines between targets, as rapidly as possible, in a seven by seven grid. There are four different conditions for the task: a numbers condition where targets go from one to forty nine (numbers), a letters condition were the targets go from A to Z followed by letters A to W with an asterisk to signify the letters as the second instance (letters), A condition where participants will alternate between numbers and letters swapping between numbers one to twenty five and letters A to X (numbers-letters) and finally a condition alternating between letters and numbers alternating between letters A to Y and numbers one and twenty four (letters-numbers). Participants will be given 20 s to make as many connections as possible on each task condition. Total number of correct connections will be recorded.
Change in verbal memory | Baseline and 24 weeks post intervention
  The Rey's auditory verbal learning test will be used to assess verbal memory. Participants will be read a list of fifteen common words five times. Immediately after each reading, they will recall as many words as possible. Next an interference list will be read containing fifteen different words, after which participants will be asked to recall the original list. In the last trial participants will be asked to recall the original list after a twenty minute delay.
Change in processing speed | Baseline and 24 weeks post intervention
  A variation on the Stroop Test performed on a laptop using Open Sesame software will be used to assess processing speed. During this task a fixation point appears on screen for 500 milliseconds followed by the presentation of the names of one of four colors blue, red, green or white. These words will be presented in four different colors again this could be either blue, red, green or white. Participants will be instructed to identify, as quickly as possible, the color of the text rather than the word displayed on screen and press a designated key on the keyboard for each of the colors. The test is comprised of 144 trials with half of trials having the text and color match and half being a non-match. Processing speed is automatically calculated by the software and is defined as the difference between the mean time taken to respond to the match and non-math trials.
Change in spatial working memory | Baseline and 24 weeks post intervention
  This task takes place on a laptop using Open Sesame software. Participants are asked to recall the spatial locations of three dots that appear in random locations on screen. The task consists on 10 practice trials followed by 60 recorded trials, with percentage of correct answers being recorded.
Change in fast walking speed | Baseline and 24 weeks post intervention
  Fast walking speed will be measured using inertial measurement sensors and results will be expressed in m/s. Participants will be asked to walk as fast as possible over 13 m. Acceleration and deceleration periods will automatically be excluded from analysis and the measure will be repeated five times with the highest value being recorded.
Change in dual task walking speed | Baseline and 24 weeks post intervention
  Dual task walking speed will be measured using inertial measurement sensors and will be expressed in m/s. This task will require participants to walk whilst counting backwards in integers of three from a randomly generated three digit number. This number will be given three seconds before the participant is prompted to start walking. No instruction will be given on prioritization of tasks and the measure will be repeated five times, with the mean gait speed being recorded.
Change in dual Task Cost | Baseline and 24 weeks post intervention
  The percentage difference between single and dual task performance calculated as = 100* (single-task score - dual-task score)/ single-task
Change in five times sit to stand | Baseline and 24 weeks post intervention
  For this task participants will start off seated on a standard chair 44 cm in height from the ground, with their arms folded across their chest and back against the chair. They will be asked to stand up fully from the chair and sit back down again five times, whilst keeping their arms in the same position. This task will be assessed by timing participants from the prompt to start until they reached a seated position on the fifth repetition.
Change in physical functioning from short form 36 questionnaire | Baseline and 24 weeks post intervention
  Participants will be asked to complete the short form 36 questionnaire. All questions are multiple choice and scores range from zero to one hundred, with a higher score indicting a greater health status. Items 3-12 are used to assess physical functioning.
Change in bodily pain from short form 36 questionnaire | Baseline and 24 weeks post intervention
  Participants will be asked to complete the short form 36 questionnaire. All questions are multiple choice and scores range from zero to one hundred, with a higher score indicting a greater health status. Items 22 and 23 are used to assess bodily pain.
Change in role limitations due to physical health problems from short form 36 questionnaire | Baseline and 24 weeks post intervention
  Participants will be asked to complete the short form 36 questionnaire. All questions are multiple choice and scores range from zero to one hundred, with a higher score indicting a greater health status. Items 13-16 are used to assess role limitations due to physical health problems.
Change in role limitations due to personal or emotional problems from short form 36 questionnaire | Baseline and 24 weeks post intervention
  Participants will be asked to complete the short form 36 questionnaire. All questions are multiple choice and scores range from zero to one hundred, with a higher score indicting a greater health status. Items 17-19 are used to assess role limitations due to personal or emotional problems.
Change in emotional well-being from short form 36 questionnaire | Baseline and 24 weeks post intervention
  Participants will be asked to complete the short form 36 questionnaire. All questions are multiple choice and scores range from zero to one hundred, with a higher score indicting a greater health status. Items 24-26, 28 and 30 are used to assess emotional well-being.
Change in social functioning from short form 36 questionnaire | Baseline and 24 weeks post intervention
  Participants will be asked to complete the short form 36 questionnaire. All questions are multiple choice and scores range from zero to one hundred, with a higher score indicting a greater health status. Items 20 and 32 are used to assess social functioning.
Change in energy/fatigue from short form 36 questionnaire | Baseline and 24 weeks post intervention
  Participants will be asked to complete the short form 36 questionnaire. All questions are multiple choice and scores range from zero to one hundred, with a higher score indicting a greater health status. Items 23, 27, 29 and 31 are used to assess energy/fatigue.
Change in general health perceptions from short form 36 questionnaire | Baseline and 24 weeks post intervention
  Participants will be asked to complete the short form 36 questionnaire. All questions are multiple choice and scores range from zero to one hundred, with a higher score indicting a greater health status. Items 1 and 33-36 are used to assess general health perceptions.

OTHER OUTCOMES:
Change in whole-blood fatty acid content | Baseline and 24 weeks post intervention
  Whole-blood fatty acid content will be analyzed from finger-prick samples from non-fasted participants.
Change in serum homocysteine | Baseline and 24 weeks post intervention
  Serum homocysteine levels will be measured by a commercially available enzyme-linked immunosorbent assay (ELISA).
Change in stride length | Baseline and 24 weeks post intervention
  Change in stride length will be recorded on each gait outcome, using inertial measurement sensors, to give an insight into which aspects of the gait cycle are driving any changes that occur.
Change in cadence | Baseline and 24 weeks post intervention
  Change in cadence will be recorded on each gait outcome, inertial measurement sensors, to give an insight into which aspects of the gait cycle are driving any changes that occur.
Change in double support phase percentage | Baseline and 24 weeks post intervention
  Change in double support phase percentage will be recorded on each gait outcome, inertial measurement sensors, to give an insight into which aspects of the gait cycle are driving any changes that occur.
Change in stride length variability | Baseline and 24 weeks post intervention
  Change in stride length variability will be recorded on each gait outcome, inertial measurement sensors, to give an insight into which aspects of the gait cycle are driving any changes that occur.
Physical activity levels | Baseline and 24 weeks post intervention
  Physical activity levels will be assessed using the previously validated community health activities program for seniors questionnaire.
Dietary energy intake | Baseline and 24 weeks post intervention
  Dietary energy intake will be assessed using a estimated three day diet diary. Diet diaries will be analyzed using nutritional composition analysis software and result expressed as kilocalories per day.
Carbohydrate intake from diet | Baseline and 24 weeks post intervention
  Carbohydrate intake will be assessed using a estimated three day diet diary. Diet diaries will be analyzed using nutritional composition analysis software and result expressed as grams per day.
Protein intake from diet | Baseline and 24 weeks post intervention
  Protein intake will be assessed using a estimated three day diet diary. Diet diaries will be analyzed using nutritional composition analysis software and result expressed as grams per day.
Fat intake from diet | Baseline and 24 weeks post intervention
  Fat intake will be assessed using a estimated three day diet diary. Diet diaries will be analyzed using nutritional composition analysis software and result expressed as grams per day.
Omega-3 polyunsaturated fatty acid intake from diet | Baseline and 24 weeks post intervention
  Omega-3 polyunsaturated fatty acid intake will be assessed using a previously validated 17 item food frequency questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Simon C Dyall, PhD, Principal Investigator — Bournemouth University; Fotini Tsofliou, PhD, Study Director — Bournemouth University
Locations (1):
- Bournemouth University, Bournemouth, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Strike SC, Carlisle A, Gibson EL, Dyall SC. A High Omega-3 Fatty Acid Multinutrient Supplement Benefits Cognition and Mobility in Older Women: A Randomized, Double-blind, Placebo-controlled Pilot Study. J Gerontol A Biol Sci Med Sci. 2016 Feb;71(2):236-42. doi: 10.1093/gerona/glv109. Epub 2015 Aug 11. PMID 26265727
- [Background] Dyall SC. Long-chain omega-3 fatty acids and the brain: a review of the independent and shared effects of EPA, DPA and DHA. Front Aging Neurosci. 2015 Apr 21;7:52. doi: 10.3389/fnagi.2015.00052. eCollection 2015. PMID 25954194
- [Background] Dyall SC. Methodological issues and inconsistencies in the field of omega-3 fatty acids research. Prostaglandins Leukot Essent Fatty Acids. 2011 Nov;85(5):281-5. doi: 10.1016/j.plefa.2011.04.009. Epub 2011 Sep 16. PMID 21925854
- [Derived] Fairbairn P, Tsofliou F, Johnson A, Dyall SC. Combining a high DHA multi-nutrient supplement with aerobic exercise: Protocol for a randomised controlled study assessing mobility and cognitive function in older women. Prostaglandins Leukot Essent Fatty Acids. 2019 Apr;143:21-30. doi: 10.1016/j.plefa.2019.04.001. Epub 2019 Apr 1. PMID 30975379